CLINICAL TRIAL: NCT06200012
Title: Multi-Level Stigma Intervention to Improve Access to Substance Use Care With Prescribing Providers in Mental Health Settings
Brief Title: Multi-Level Stigma Intervention for Mental Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: University of New Mexico (Other); Loyola University Chicago (Other); LifeStance Health (Unknown)
Responsible Party: Principal Investigator, Erin F. Madden, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UG1DA049468 CTN-00137; UG1DA049468 (NIH)
Record Dates: First submitted 2023-11-30; First posted 2024-01-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Social Stigma; Substance Use Disorders; Mental Disorder
MeSH Terms: conditions — Social Stigma; Substance-Related Disorders; Mental Disorders

STUDY DESIGN:
Masking Description: Providers in the experimental and control arms are are not masked. Providers in the experimental arm have a policy at their clinic change, and they are aware of the policy change. The control arm does not implement the policy change, but may be aware of the policy change in the other arm. Both arms receive an educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control arm: educational training only (Active Comparator): This arm received only an educational training for mental health professionals about substance use-related stigma
  Interventions: Behavioral: Single-level stigma reduction intervention: educational training
- Experimental arm: educational training plus a policy change for controlled substance agreements (Experimental): This arm received both 1) an educational training for mental health professionals about substance use-related stigma; and 2) a policy change that replaced the standard LifeStance Health system's "controlled substance agreement" (CSA) with a new agreement integrating principles of shared decision-making and offering prescribers a communication tool with suggestions for how to implement principles of shared decision-making and patient centered care in their use of the new CSA
  Interventions: Behavioral: Multi-level stigma reduction intervention: educational training plus controlled substance agreement policy change

INTERVENTIONS:
Behavioral: Multi-level stigma reduction intervention: educational training plus controlled substance agreement policy change — Pairing a professional training targeting known attitudinal and knowledge drivers of substance use stigma with a policy altering potentially stigmatizing features of controlled substance agreements.
  Arms: Experimental arm: educational training plus a policy change for controlled substance agreements
Behavioral: Single-level stigma reduction intervention: educational training — A professional training targeting known attitudinal and knowledge drivers of substance use stigma
  Arms: Control arm: educational training only

SUMMARY:
This cluster randomized trial develops and pilot tests a multi-level substance use stigma intervention that leverages organizational policy and professional education to address structural and professional drivers of stigma in outpatient mental health (MH) services. The investigators will generate preliminary data to determine whether adding an organizational policy to a professional stigma training may reduce measures of provider-based stigma towards substance use and improve care quality and patient outcomes to a greater degree than simply conducting training alone. The investigators hypothesize that providers at a MH site implementing an organizational policy change in addition to providing professional training will demonstrate greater improvement to health services for people who use drugs compared to a site where providers receive training alone.

DETAILED DESCRIPTION:
Substance use is commonly stigmatized, even in health settings. Stigma toward people who use drugs (PWUD) arises from multiple sources, including policies and individuals who carry out policies ("structural stigma") and health professionals ("provider-based stigma"). This study seeks to answer the question of whether addressing organizational-level structural stigma toward PWUD enhances the behavioral effects of stigma training among professionals providing mental health (MH) services.

This study will have two intervention groups: A MH clinic where the providers receive only the educational intervention and a MH clinic where the providers receive both the educational intervention and an organizational policy change. The investigators hypothesize that providers at a MH site implementing an organizational policy change in addition to providing professional training will demonstrate greater improvement to health services for PWUD compared to a site where providers receive training alone.

Only a small body of research develops and evaluates interventions seeking to reduce structural and provider-based stigma toward PWUD in healthcare settings or investigates the impact of such interventions on provision of evidence-based interventions like substance use disorder (SUD) pharmacotherapy. Little is known about substance use stigma in MH settings in particular, although some research suggests psychiatrist stigma toward dual diagnosis patients is greater than toward patients with either a SUD or MH diagnosis alone. Extant studies on stigma toward PWUD in healthcare found educational interventions incorporating critical reflection techniques and contact with PWUD significantly reduced provider-based stigma. But most provider-based stigma intervention studies have two major weaknesses: 1) failing to address structural drivers of stigma, such as organizational policies motivating attitudes and behaviors, and 2) falling short of practical application because they largely focus on professional attitudes without measuring changes to service provision. The investigators propose to pilot test a multi-level stigma intervention that leverages what existing research suggests works in professional stigma education, and adds a novel component of organizational policy change within a MH clinic. Because so little research exists on organizational-level stigma interventions, the investigators will use an inductive approach to identify a promising feasible policy that may reduce stigma toward PWUD. Our pilot testing will assess the extent to which combining interventions that modify structural/organizational and individual/professional-level drivers of stigma in outpatient MH services may improve not only attitudes but also health service provision to PWUD.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the inclusion criteria in order to be eligible to participate in the study.

1. Site inclusion:

   * The sites will be selected using convenience sampling.
   * The inclusion criterion will be sites with at least 4 providers.
2. Provider inclusion:

   * Providers at participating sites will also be recruited using convenience sampling.
   * Any psychiatrists or psychiatric NPs are eligible to participate as long as they are employed at the participating LSH site.
3. Patient EHR inclusion:

   * All new patients entering mental health services during the 3-months prior and 3- months after the intervention will be included in the EHR data sample to assess whether substance use was addressed during their first visit and subsequent 3-month retention in care.
   * Existing and new patients with alcohol use disorder (AUD)/opioid use disorder (OUD) will be identified through the EHR to assess pharmacotherapy initiation.
4. Patient survey inclusion:

   * Half of the survey sample (n=20) will include patients without a substance use disorder (SUD) documented in their chart at the time of data collection
   * The other half of the survey sample (n=20) will include patients who do have an ICD-10 code for SUD in their chart.
   * Patient stratification rationale: the intention is to compare experiences and perceptions of stigma among patients who have SUD noted in their EHR and those who do not. This is also to assess stigma among patients who may not have their substance use addressed during a MH visit but who have substance use related health risks and substance use disorders (assessed through the ASSIST questionnaire).

Exclusion Criteria:

All individuals meeting any of the exclusion criteria will be excluded from study participation.

1. Provider exclusion:

   * Providers may be excluded if they were not employed by LSH and seeing patients for the past three months at the time of enrollment.
2. Patient exclusion:

   * Patients may be excluded from the SUD-stratified portion of the survey sample if their SUD diagnosis is only for a tobacco use disorder.
   * Patients may also be excluded if they are unable or unwilling to give written informed consent.
   * Patients who are currently in jail, prison or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Number of patients where substance use was addressed during a MH visit among new intakes and documented in EHR | 3-months prior to intervention vs. 3-months after intervention
  Identified ICD-10s or notes among participating providers in electronic health records (EHR)
Number of patients in the provider panel (new or old) diagnosed with OUD or AUD who initiated OUD or AUD pharmacotherapy | 3-months prior to intervention vs. 3-months after intervention
  Whether pharmacotherapy for opioid use disorders (OUD) or alcohol use disorders (AUD) was initiated for patients with ICD-10s for OUD or AUD, as indicated in electronic health records (EHR)
Three-month retention in MH services for new patients whose EHR indicate substance use or SUD | 3-months prior to intervention vs. 3-months after intervention
  Measured as any return visit for mental health (MH) services, as documented in electronic health records (EHR) for patients with ICD-10s for substance use disorders (SUD) or any indication of substance use in provider notes

SECONDARY OUTCOMES:
Training intervention feasibility | up to 14 days after training
  Assessed among professionals in training using Feasibility of Intervention Measure (FIM) in post-training surveys
Training intervention acceptability | up to 14 days after training
  Assessed among professionals in training using Acceptability of Intervention Measure (AIM) in post-training surveys
Training intervention appropriateness | up to 14 days after training
  Assessed among professionals in training using Intervention Appropriateness Measure (IAM) in post-training surveys
Professional Stigma measured with Social Distance Scale (SDS) | up to 14 days before training, up to 14 days after training, and 6-weeks after training
  Measures willingness to have several kinds of social relationships among professionals in training, and adapted for three populations: relationships with people who actively use drugs, with people who used to use drugs, and with people treated with opioid agonist treatment. Assessed in longitudinal surveys (within 14 days pre-training, within 14 days post-training, and 6-weeks post-training). Lower score indicates greater stigma, min=12 and max=60.
Professional Stigma measured with Medical Condition Regard Scale (MCRS) | up to 14 days before training, up to 14 days after training, and 6-weeks after training
  Measures endorsed provider-based stigma toward patients with a specific diagnosis among professionals in training. Assessed in longitudinal surveys (within 14 days pre-training, within 14 days post-training, and 6-weeks post-training). Lower score indicates greater stigma, min=7 and max=35.
Professional Stigma measured with Perceived Dangerousness Scale | up to 14 days before training, up to 14 days after training, and 6-weeks after training
  Measures perceptions of the dangerousness of a stigmatized group among professionals in training. Assessed in longitudinal surveys (within 14 days pre-training, within 14 days post-training, and 6-weeks post-training). Lower score indicates greater stigma, min=5 and max=25.
Patient-reported stigma measured with Internalized Stigma of Mental Illness Inventory (ISMI) | 6-week post-training survey
  This measure is for patients and includes questions about anticipated stigma and internalized/self-stigma. This will be asked of a stratified random sample of patients of participating providers (n=20 with a SUD and n=20 not diagnosed with an SUD). Lower score indicates less stigma, min=29 and max=116.

CONTACTS AND LOCATIONS:
Locations (1):
- LifeStance Health, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary data for this study will be available to the public in the NIDA data repository, per NIDA CTN policy.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of primary outcomes analysis